CLINICAL TRIAL: NCT02453659
Title: Distress Tolerance Treatment for Weight Concern in Smoking Cessation Among Women
Brief Title: Women Engaging in Quitting Smoking Together
Acronym: WE QUIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 215114; K23DA035288 (NIH)
Record Dates: First submitted 2015-05-21; First posted 2015-05-25 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Distress Tolerance Treatment for Weight Concern (DT-W) (Experimental): DT-W is delivered over a 9 week period with 1 1-hr individual session during week 1, 8 weekly 1.5-hr group counseling sessions during weeks 2-9, and 1 20-minute individual telephone session during week 4. Session content includes distress tolerance intervention for weight concern plus standard behavioral smoking cessation treatment. Participants also receive 8 weeks of nicotine patch.
  Interventions: Behavioral: Distress Tolerance Treatment for Weight Concern (DT-W); Behavioral: Smoking Cessation counseling; Drug: Transdermal Nicotine Patch
- Health Education (HE) (Active Comparator): HE is delivered over a 9 week period with 1 1-hr individual session during week 1, 8 weekly 1.5-hr group counseling sessions during weeks 2-9, and 1 20-minute individual telephone session during week 4. Session content includes smoking health education program plus standard behavioral smoking cessation treatment. Participants also receive 8 weeks of nicotine patch.
  Interventions: Behavioral: Health Education (HE); Behavioral: Smoking Cessation counseling; Drug: Transdermal Nicotine Patch

INTERVENTIONS:
Behavioral: Distress Tolerance Treatment for Weight Concern (DT-W)
  Arms: Distress Tolerance Treatment for Weight Concern (DT-W)
Behavioral: Health Education (HE)
  Arms: Health Education (HE)
Behavioral: Smoking Cessation counseling
Drug: Transdermal Nicotine Patch

SUMMARY:
The long-term goal of this program of research is to develop and disseminate an efficacious, group-based distress tolerance treatment for weight concern (DT-W) that will significantly increase smoking cessation rates among women. The objective of this project is to conduct a preliminary randomized controlled trial (RCT) (N = 60) comparing DT-W to a Health Education (HE) comparison intervention, in which both groups also receive standard behavioral smoking cessation treatment (ST) including counseling and transdermal nicotine patch (TNP), and examine potential mechanisms that may underlie the efficacy of DT-W in improving smoking outcomes at 1-, 3-, and 6-month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

female

* at least 18 years of age
* smoke 5 or more cigarettes per day
* daily smoker for at least the past year
* report motivation to quit smoking in the next month of at least 5 on a 10 point scale
* report concern of at least 50 on at least one of two 100 point scales assessing weight concern
* able to travel to study location for study appointments

Exclusion Criteria:

* current use of other smoking cessation or weight loss therapies
* current use of other tobacco products at least weekly
* diagnosis or treatment for non-nicotine substance use disorder with substance use during the past 6 months
* lifetime diagnosis or treatment of eating disorder, bipolar disorder, schizophrenia, or schizoaffective disorder
* score above established cut-offs on self-report screening measures of depressive symptomology, eating disorder symptomology, alcohol use disorder, or drug use disorder
* current suicidality or homicidality
* medical condition that is a contraindication for the use of transdermal nicotine patch
* lives at same address as current or past participant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Point prevalence abstinence from smoking: percentage of participants in each treatment group who report abstinence from smoking for the 7 days prior to each follow-up assessment | 6 months post-quit date
  The investigators will compare the percentage of participants in each treatment group who report abstinence from smoking for the 7 days prior to each follow-up assessment (1-, 3-, and 6-months post-quit date).

CONTACTS AND LOCATIONS:
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Hartmann-Boyce J, Theodoulou A, Farley A, Hajek P, Lycett D, Jones LL, Kudlek L, Heath L, Hajizadeh A, Schenkels M, Aveyard P. Interventions for preventing weight gain after smoking cessation. Cochrane Database Syst Rev. 2021 Oct 6;10(10):CD006219. doi: 10.1002/14651858.CD006219.pub4. PMID 34611902